CLINICAL TRIAL: NCT00089258
Title: Phase II Study of Anti-GD2 3F8 Antibody and Biologic Response Modifiers for High-risk Neuroblastoma
Brief Title: Biological Therapy in Treating Patients With Neuroblastoma That Has Not Responded to Previous Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: 04-050; MSKCC-04050
Record Dates: First submitted 2004-08-04; First posted 2004-08-05 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2013-01

CONDITIONS: Neuroblastoma
Keywords: localized unresectable neuroblastoma; disseminated neuroblastoma; regional neuroblastoma; stage 4S neuroblastoma; recurrent neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — beta-Glucans; humanized 3F8 anti-GD2 monoclonal antibody; sargramostim; Isotretinoin

INTERVENTIONS:
Biological: beta-glucan
Biological: monoclonal antibody 3F8
Biological: sargramostim
Drug: isotretinoin

SUMMARY:
RATIONALE: Monoclonal antibodies, such as monoclonal antibody 3F8, can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Beta-glucan, isotretinoin, and sargramostim may increase the effectiveness of monoclonal antibody 3F8 by making tumor cells more sensitive to the monoclonal antibody. Combining different types of biological therapy may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving beta-glucan, isotretinoin, and sargramostim together with monoclonal antibody 3F8 works in treating patients with neuroblastoma that has not responded to previous treatment.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of beta-glucan, isotretinoin, and sargramostim (GM-CSF) in enhancing monoclonal antibody 3F8-mediated ablation in patients with high-risk refractory neuroblastoma.
* Determine the antitumor activity of this regimen, in terms of assessing disease status in the bone marrow by real-time quantitative reverse transcription polymerase chain reaction, in these patients.
* Determine the toxicity of this regimen in these patients.

OUTLINE: This is an open-label study. Patients are stratified according to refractory disease (primary refractory [never had disease progression or disease recurrence] vs secondary refractory [recurrent disease that did not respond completely to reinduction therapy]).

* Courses 1 and 2: Patients receive sargramostim (GM-CSF) subcutaneously once daily on days -5 to 11. Patients also receive oral beta-glucan once daily on days -2 to 11 and monoclonal antibody (MOAB) 3F8 IV over 30-90 minutes on days 0-4 and 7-11.
* Courses 3 and 4: Patients receive GM-CSF, beta-glucan, and MOAB 3F8 as above. Patients also receive oral isotretinoin twice daily on days -2 to 11.

Treatment repeats every 2-4 weeks for 4 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years.

PROJECTED ACCRUAL: A total of 27-74 patients (10-33 for stratum 1 and 17-41 for stratum 2) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of neuroblastoma, as defined by 1 of the following:

  * Histologically confirmed disease
  * Bone marrow metastases plus high urine catecholamines
* High-risk disease meeting 1 of the following stage criteria:

  * Stage IV, with 1 of the following:

    * Any age with MYCN amplification
    * > 18 months of age without MYCN amplification
  * Stage III, with both of the following:

    * Any age with MYCN amplification
    * Unresectable disease
  * Stage 4S with MYCN amplification
* Measurable or evaluable soft tissue disease
* Relapsed disease resistant to standard induction chemotherapy and salvage therapy

PATIENT CHARACTERISTICS:

Age

* Any age

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* No severe hepatic toxicity ≥ grade 3

Renal

* No severe renal toxicity ≥ grade 3

Cardiovascular

* No severe cardiac toxicity ≥ grade 3

Pulmonary

* No severe pulmonary toxicity ≥ grade 3

Other

* Not pregnant
* Negative pregnancy test
* No severe neurologic toxicity ≥ grade 3
* No severe gastrointestinal toxicity ≥ grade 3
* No other severe major organ dysfunction except ototoxicity
* No history of allergy to mouse proteins
* No active life-threatening infection
* No human anti-mouse antibody titer > 1,000 ELISA units/mL

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2004-07; Primary Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Disease response as assessed by PT-PC at the end of 4 courses

CONTACTS AND LOCATIONS:
Overall Officials: Nai-Kong V. Cheung, MD, PhD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States